CLINICAL TRIAL: NCT05223426
Title: A Multicenter Randomized Single-blinded Clinical Trial to Investigate the Effects of a Home-based Cognitive Training for individualS Affected bY chroNic heArt Failure: an Individualized Program to increaSE Cognitive Functions
Brief Title: Effects of Individualized Cognitive Training on Cognition in Heart Failure
Acronym: SYNAPSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Louis Bherer (Other)
Collaborators: The Montreal Health Innovations Coordinating Center (MHICC) (Other)
Responsible Party: Sponsor-Investigator, Louis Bherer, Associate scientific director, Direction of prevention, Montreal heart Institute, Montreal Heart Institute
Organization: Montreal Heart Institute (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: MP-33-2022-2981
Record Dates: First submitted 2021-09-29; First posted 2022-02-04 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure
Keywords: Heart failure; Cognition; Individualized cognitive training; Home-based intervention; Remote monitoring
MeSH Terms: conditions — Heart Failure | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single blind masking: the research personnel performing the outcome assessments at baseline, between the intervention (two months) and after the intervention (four months) will be blinded to groups' intervention order. Participants will be aware of the order in which they receive the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive training followed by usual care (Experimental): Usual care and cognitive training for 6 weeks, followed by usual care (only) for 6 weeks.
  Interventions: Other: Cognitive training; Other: Usual Care
- Usual care followed by cognitive training (Experimental): Usual care (only) for 6 weeks, followed by cognitive training and usual care for 6 weeks.
  Interventions: Other: Cognitive training; Other: Usual Care

INTERVENTIONS:
Other: Cognitive training — A cognitive training program will be individually developed for each participant based on baseline neuropsychological tests. It will include: Computerized cognitive training: this training include: the Dual-Task, the Stroop and the N-Back task. The tasks are accompanied by feedback based on the participant's responses (e.g., progress graph, feedback, etc.). In order to promote participants' learning, the level of difficulty of the tasks increased as training sessions progressed. Two sets of stimuli will be used to maximize the generalization of learning. Memory training: This training is adapted from the MEMO+ training program (Belleville et al., 2018). These sessions, also home-based, will be done through online video and are covering a variety of topics: memory (normal aging, mnemonic strategies), attention, aging, etc. Each week, participants will be asked to complete the equivalent of 6 training sessions of 15 minutes each, for a total of 1h30 per week.
Other: Usual Care — Participants will be asked to continue the care and follow-up as usually planned with the attending cardiologist. Apart from weekly follow-ups with the research team member, no changes will be made to the participant's medical care.

SUMMARY:
The SYNAPSE trial is designed to study the effects of an individualized home-based cognitive training program on cognitive functions in heart-failure patients.

DETAILED DESCRIPTION:
The purpose of the SYNAPSE study is to evaluate the effects of an individualized home-based training program aimed to improve cognitive functions and well-being in heart failure patients. Heart failure is characterized by the inability of the heart to pump blood efficiently through the body. Nearly half of patients with heart failure present with cognitive deficits. Memory and executive functions that allow us to perform complex tasks are mainly affected. These cognitive deficits are linked to an increased risk of hospitalization and mortality, in addition to decreasing patients' well-being and ability to care for themselves. Although rehabilitation programs that include physical activity and counseling help reduce heart and brain health risks, these programs are unpopular. Among the few who enroll, between 24% and 50% drop out before the completion of the program. Offering alternative options such as cognitive training would help to reach this proportion of patients. The literature has shown that cognitive training is effective in preventing or reducing cognitive deficits in older adults with or without cognitive loss. Although still understudied in patients with heart failure, a better understanding of the association between heart failure and changes in cognition would allow better adaptation of patient care to their situations and needs.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 50 or older
* Have access to Internet
* Have access to a computer or a tablet;
* Have the ability to perform cognitive training;
* Have the ability to read, understand and consent to the informed consent form;
* Have chronic heart failure on tolerated therapy for at least two months;
* Without limitation of physical activity to severe limitation of physical activity (i.e. NYHA class I, class II, class III OR class IV).

Exclusion Criteria:

* Acute cardiovascular event 1 month before randomization;
* Cardiovascular procedure scheduled within 3 months;
* Uncontrolled diabetes or untreated thyroid dysfunction;
* Current or recent malignancy with a life expectancy of less than 1 year;
* Neurological disease;
* Chronic hemodialysis or peritoneal dialysis.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Changes in performance on trained computerized cognitive tasks | Before and after the 6 weeks of interventions
  Trained version of computerized dual-task, modified stroop and n-back tasks
  Reaction time (ms)
Changes in performance on trained computerized cognitive tasks | Before and after the 6 weeks of interventions
  Trained version of computerized dual-task, modified stroop and n-back tasks
  Accuracy (%)
Changes in performance on transfer computerized cognitive tasks | Before and after the 6 weeks of interventions
  Transfer version of computerized dual-task, modified stroop and n-back tasks
  Reaction time (ms)
Changes in performance on transfer computerized cognitive tasks | Before and after the 6 weeks of interventions
  Transfer version of computerized dual-task, modified stroop and n-back tasks
  Accuracy (%)

SECONDARY OUTCOMES:
Change in general cognitive functioning | Before and after the 6 weeks of interventions
  Remote version of the Montreal Cognitive Assessment. (0-28 score, with a higher score indicating a better cognitive functioning.)
Changes in performance on neuropsychological tests | Before and after the 6 weeks of interventions
  Remote version of validated neuropsychological test
  Memory capacity
  -Rey Auditory Verbal Learning Test
  (z-score change)
Changes in performance on neuropsychological tests | Before and after the 6 weeks of interventions
  Remote version of validated neuropsychological test
  Processing speed
  -Trail making test Part A
  (z-score change)
Changes in performance on neuropsychological tests | Before and after the 6 weeks of interventions
  Remote version of validated neuropsychological test
  Executive functions
  * Trail making test Part B
  * Verbal fluency test
  * Digit span test
    (z-score change)
Change in quality of life | Before and after the 6 weeks of interventions
  36-Items Short form health Survey (SF-36) (Score ranges from 0-100, with a higher score indicating more favorable health status.)
Change in self-care behavior | Before and after the 6 weeks of interventions
  European Heart-Failure Self-care Behavior Scale-9 (EHFsB-9) (The minimal score is 9 while the maximal score is 45. The higher the score, the less the patient performs self-care behaviors.)

OTHER OUTCOMES:
Change in depressive symptomatology | Before and after the 6 weeks of interventions
  Patient Health Questionnaire (PHQ-9) (Score ranges from 0 to 27, with a higher score indicating a more severe depression state.)
Change in anxiety | Before and after the 6 weeks of interventions
  General Anxiety Disorder questionnaire (GAD-7) (Total score ranges from 0 to 21, with an increasing score on the scale is indicating a worse anxiety state.)
Change in perceived stress | Before and after the 6 weeks of interventions
  Perceived Stress Scale questionnaire (PSS-10) (Score ranges from 0-40, with a higher score indicating a worse sleep quality)
Change in quality of sleep | Before and after the 6 weeks of interventions
  Pittsburgh Sleep Quality Index questionnaire (PSQI) (19 self-assessment questions are grouped into seven components. The scores for the seven components are summed to give an overall score that ranges from 0 to 21 points, with "0" indicating no difficulty and "21" indicating severe difficulty in all components. A score higher than 5 indicates problematic sleep in one or more components)
Change in Risk of sleep apnea | Before and after the 6 weeks of interventions
  Berlin Questionnaire (Participants are classified into a high or a low risk of sleep apnea based their responses to the individual items and their overall scores in the symptom categories. A High Risk represent 2 or more categories where the score is positive. A low risk represents 1 or no category where the score is positive.)
Change in self-reported physical activity | Before and after the 6 weeks of interventions
  Physical Activity Scale for the Elderly Questionnaire (PASE) (The overall score ranges from 0 to 400, with a higher score indicating a better level of physical activity)
Change in Walking test speed | Before and after the 6 weeks of interventions
  4-meter walking test (m/s)
Change in functional mobility | Before and after the 6 weeks of interventions
  Timed up and Go test (s)
Change in balance performance | Before and after the 6 weeks of interventions
  Timed one-leg standing test (s)
Change in lower limb muscles strength | Before and after the 6 weeks of interventions
  Timed Sit-to-Stand test (s)
Cognitive Reserve | Baseline
  Rami and colleagues' cognitive reserve questionnaire (Scale ranges from 0-26, with a higher score indicating a greater cognitive reserve)
Self-reported masculinity and femininity traits | Baseline
  Short Form BEM Sex-Role Inventory questionnaire (30 items questionnaire with 10 items assessing the femininity traits, 10 items assessing the masculinity traits and 10 items neutral, not scored. Two scores, rage from 10-70, are calculated for femininity and masculinity, respectively. A higher score is indicating a higher trait.)
Dietary patterns | Baseline
  Short Diet Questionnaire (Score ranges from 15-45 points, with a score between 15-29 categorized as unhealthy, 30-37 as somewhat unhealthy and 38 or more as a healthy diet.)

CONTACTS AND LOCATIONS:
Overall Officials: Louis Bherer, PhD, Principal Investigator — Montreal Heart Institute
Locations (2):
- Canada (2):
  - Preventive medicine and physical activity center (centre EPIC), Montreal heart Institute, Montreal, Quebec
  - Centre de recherche du centre Hospitalier de l'Université de Montréal (CRCHUM), Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Turk-Adawi KI, Oldridge NB, Tarima SS, Stason WB, Shepard DS. Cardiac rehabilitation patient and organizational factors: what keeps patients in programs? J Am Heart Assoc. 2013 Oct 21;2(5):e000418. doi: 10.1161/JAHA.113.000418. PMID 24145743
- [Background] Resurreccion DM, Moreno-Peral P, Gomez-Herranz M, Rubio-Valera M, Pastor L, Caldas de Almeida JM, Motrico E. Factors associated with non-participation in and dropout from cardiac rehabilitation programmes: a systematic review of prospective cohort studies. Eur J Cardiovasc Nurs. 2019 Jan;18(1):38-47. doi: 10.1177/1474515118783157. Epub 2018 Jun 18. PMID 29909641
- [Background] Rego MLM, Cabral DAR, Fontes EB. Cognitive Deficit in Heart Failure and the Benefits of Aerobic Physical Activity. Arq Bras Cardiol. 2018 Jan;110(1):91-94. doi: 10.5935/abc.20180002. PMID 29538528
- [Background] Leto L, Feola M. Cognitive impairment in heart failure patients. J Geriatr Cardiol. 2014 Dec;11(4):316-28. doi: 10.11909/j.issn.1671-5411.2014.04.007. PMID 25593581
- [Background] Hawkins MA, Schaefer JT, Gunstad J, Dolansky MA, Redle JD, Josephson R, Moore SM, Hughes JW. What is your patient's cognitive profile? Three distinct subgroups of cognitive function in persons with heart failure. Appl Nurs Res. 2015 May;28(2):186-91. doi: 10.1016/j.apnr.2014.10.005. Epub 2014 Oct 31. PMID 25510559
- [Background] Doehner W. Dementia and the heart failure patient. Eur Heart J Suppl. 2019 Dec;21(Suppl L):L28-L31. doi: 10.1093/eurheartj/suz242. Epub 2019 Dec 23. PMID 31885510
- [Background] Dodson JA, Chaudhry SI. Geriatric conditions in heart failure. Curr Cardiovasc Risk Rep. 2012 Oct;6(5):404-410. doi: 10.1007/s12170-012-0259-8. PMID 23997843
- [Background] Dickson VV, Tkacs N, Riegel B. Cognitive influences on self-care decision making in persons with heart failure. Am Heart J. 2007 Sep;154(3):424-31. doi: 10.1016/j.ahj.2007.04.058. PMID 17719284
- [Background] de Tournay-Jette E, Dupuis G, Denault A, Cartier R, Bherer L. The benefits of cognitive training after a coronary artery bypass graft surgery. J Behav Med. 2012 Oct;35(5):557-68. doi: 10.1007/s10865-011-9384-y. Epub 2011 Nov 9. PMID 22068879
- [Background] Cannon JA, Moffitt P, Perez-Moreno AC, Walters MR, Broomfield NM, McMurray JJV, Quinn TJ. Cognitive Impairment and Heart Failure: Systematic Review and Meta-Analysis. J Card Fail. 2017 Jun;23(6):464-475. doi: 10.1016/j.cardfail.2017.04.007. Epub 2017 Apr 19. PMID 28433667
- [Background] Belleville S, Hudon C, Bier N, Brodeur C, Gilbert B, Grenier S, Ouellet MC, Viscogliosi C, Gauthier S. MEMO+: Efficacy, Durability and Effect of Cognitive Training and Psychosocial Intervention in Individuals with Mild Cognitive Impairment. J Am Geriatr Soc. 2018 Apr;66(4):655-663. doi: 10.1111/jgs.15192. Epub 2018 Jan 4. PMID 29313875
- [Background] Kua ZJ, Valenzuela M, Dong Y. Can Computerized Cognitive Training Improve Cognition in Patients With Heart Failure?: A Review. J Cardiovasc Nurs. 2019 Mar/Apr;34(2):E19-E27. doi: 10.1097/JCN.0000000000000558. PMID 30585868
- [Background] Bherer L. Cognitive plasticity in older adults: effects of cognitive training and physical exercise. Ann N Y Acad Sci. 2015 Mar;1337:1-6. doi: 10.1111/nyas.12682. PMID 25773610
- [Background] Lampit A, Hallock H, Valenzuela M. Computerized cognitive training in cognitively healthy older adults: a systematic review and meta-analysis of effect modifiers. PLoS Med. 2014 Nov 18;11(11):e1001756. doi: 10.1371/journal.pmed.1001756. eCollection 2014 Nov. PMID 25405755
- [Background] Lussier M, Gagnon C, Bherer L. An investigation of response and stimulus modality transfer effects after dual-task training in younger and older. Front Hum Neurosci. 2012 May 18;6:129. doi: 10.3389/fnhum.2012.00129. eCollection 2012. PMID 22629239
- [Background] Pendlebury ST, Welch SJ, Cuthbertson FC, Mariz J, Mehta Z, Rothwell PM. Telephone assessment of cognition after transient ischemic attack and stroke: modified telephone interview of cognitive status and telephone Montreal Cognitive Assessment versus face-to-face Montreal Cognitive Assessment and neuropsychological battery. Stroke. 2013 Jan;44(1):227-9. doi: 10.1161/STROKEAHA.112.673384. Epub 2012 Nov 8. PMID 23138443
- [Derived] Blanchette CA, Besnier F, Dupuy EG, Gagnon C, Vincent T, Rouleau JL, Bouabdallaoui N, Grau JI, Racine N, Tournoux F, Apullan FJ, Vitali P, Belleville S, Bherer L. A multicenter randomized single-blinded clinical trial to investigate the effects of an individualized home-based cognitive training program in patients with chronic heart failure: the SYNAPSE protocol. Trials. 2025 Nov 17;26(1):511. doi: 10.1186/s13063-025-09193-y. PMID 41250150